CLINICAL TRIAL: NCT05516342
Title: LEAD IT! An App to Enable Persons With Early Stage Dementia to Lead Group Activities for Their Peers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopeful Aging (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AG059443; NCT04899973 (obsolete NCT alias)
Record Dates: First submitted 2022-08-10; First posted 2022-08-25 (Actual); Results first posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-05

CONDITIONS: Dementia, Vascular; Alzheimer Disease; Dementia, Mixed
Keywords: psychosocial; social; non-pharmacological intervention
MeSH Terms: conditions — Dementia, Vascular; Alzheimer Disease; Mixed Dementias

STUDY DESIGN:
Intervention Model Description: Two quasi-experiments will be conducted. Experiment #1 will test the Beta 1 Version of the app with 24 PWD and use a pre-post design. Experiment #1's goal is to examine and improve new activities and to make final changes to the overall app structure. Experiment #2, which will test Beta 2, will be a cluster randomized trial (CRT), consisting of pre- and post-intervention measurements of two nonequivalent groups: a Treatment Group (TG)-i.e. 48 PWD who receive the intervention - and a Control Group (CG)- i.e., 48 PWD receiving standard programming / care. Since Experiment #2 will occur after all tweaking is complete, it will represent the definitive trial of LEAD IT!'s proximal and distal effects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Experimental, LEAD IT! Programming (Experimental): Participants in the Experimental / LEAD IT! arm will take part in LEAD IT! programming for 18 weeks. The programming will occur twice per week, for a total of 36 sessions.
  Interventions: Behavioral: LEAD IT! Programming
- No Intervention: Control, Standard Care / Programming (No Intervention): Participants in the Control arm will receive standard care / programming.

INTERVENTIONS:
Behavioral: LEAD IT! Programming — LEAD IT! is an intervention that enables persons with dementia to lead activities for their peers. The activities take place on tablets.
  Arms: Experimental: Experimental, LEAD IT! Programming

SUMMARY:
The proposed Phase 2 project will involve the further development and evaluation of LEAD IT!, which is a tablet-based app designed to enable persons with dementia to lead activities for their peers (i.e., other persons with dementia). The study will examine the clinical outcomes of long-term use of the app by both Resident Leaders (RLs) and Resident Players (RPs).

The Specific Aims of the proposed Phase 2 project are to:

1. Develop improved Beta 1 and Beta 2 Versions of LEAD IT! with sufficient content to facilitate six activities twice per week for 4.5 months.
2. Examine the extent to which RLs are able to serve as leaders while using LEAD IT!
3. Examine the effects of resident-led LEAD IT! programming on RPs.
4. Examine PWD and staff satisfaction with LEAD IT!

DETAILED DESCRIPTION:
he proposed Phase 2 project will involve the further development and evaluation of LEAD IT!, as well as examine the clinical outcomes of long-term use of the app by both RLs and RPs.

The Specific Aims of the proposed Phase 2 project are to:

1. Develop improved Beta 1 and Beta 2 Versions of LEAD IT! with sufficient content to facilitate six activities twice per week for 4.5 months. During Months 1-7, the Beta 1 version of the app will be created by the study's Development Team (DT). During Months 13-15, the DT will create an improved Beta 2 version, based on lessons learned in Beta 1 testing.
2. Examine the extent to which RLs are able to serve as leaders while using LEAD IT! During all intervention sessions, researchers will track the extent to which each RL follows key steps involved in leading each activity. RLs will be considered successful if they follow the steps 80% of the time and require less staff assistance on less than 20% of steps.
3. Examine the effects of resident-led LEAD IT! programming on RPs. Two quasi-experiments will be conducted. Experiment #1, which will test the Beta 1 version of LEAD IT!, will use a pre-post design. Proximal (immediate) effects will be assessed by examining RP's levels of engagement/affect during baseline (standard) activities and again during LEAD IT! activities. It is hypothesized that LEAD IT! will result in higher quality engagement than baseline activities. Experiment #2, which will test the Beta 2 version of the app, will be a cluster randomized trial (CRT), consisting of pre- and post-intervention measurements of a Treatment Group (TG)-which will consist of PWD who receive the intervention - and a Control Group (CG) - which will consist of PWD who receive standard programming / care. Since Experiment #2 will occur after all improvements to the app have been made, it will represent the definitive trial of the LEAD IT! app's impact on PWD. For proximal (immediate) measures, it is anticipated that there will be a Group x Time interaction effect, with TG participants exhibiting significantly greater increases in positive forms of engagement, as compared to CG participants. For distal measures, it is anticipated that there will be a Group x Time interaction effect, with TG participants exhibiting significantly greater increases in quality of life (based upon the DEMQOL) at treatment, as compared to CG participants.
4. Examine PWD and staff satisfaction with LEAD IT! This will be achieved by eliciting feedback from PWD and staff members. PWD and staff members will be considered "highly satisfied" with the app if 85% are satisfied with the app.

ELIGIBILITY:
Inclusion Criteria for Persons with Dementia

* Must reside in an Assisted Living Facility or NH
* Must be at least 65 years old
* Must speak and read English
* Must have a clinical diagnosis of dementia (any type).
* Resident-players must score at least five on the Mini-Mental State Examination (MMSE)
* Resident-leaders must score at least 13 on the MMSE
* Resident-leaders must possess at least 70% of the characteristics of successful leaders, based upon the I'm Still Here Skills Inventory, Short Edition, Modified

Exclusion Criteria for Persons with Dementia -the person shows signs of rapid cognitive decline or physical deterioration over the last six months, as evidenced by medical records.

Inclusion Criteria for Staff

* Must be at least 18 years old
* Must speak English

Exclusion Criteria for Staff

-n/a

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2023-06-11 (Actual); Study Completion 2023-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Skrajner, MA, Principal Investigator — Hearthstone
Locations (1):
- The Hearthstone Institute, LLC, Winchester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Long-Term Care Communities
Groups:
- Persons With Dementia, Experimental (LEAD IT! Programming): Participants in the Experimental / LEAD IT! arm will take part in LEAD IT! programming for 3 months. Participants were invited to participate in LEAD IT! programming twice per week. LEAD IT! Programming: LEAD IT! is an intervention that enables persons with dementia to lead activities for their peers. The activities take place on tablets.
- Persons With Dementia, Control (Standard Care / Activity Programming): Participants in the Control arm will receive standard care / programming.
Period: Baseline
Arm/Group | Persons With Dementia, Experimental (LEAD IT! Programming) | Persons With Dementia, Control (Standard Care / Activity Programming)
Started | 54; 5 Long-Term Care Communities | 41; 4 Long-Term Care Communities
Completed | 54; 5 Long-Term Care Communities | 41; 4 Long-Term Care Communities
Not Completed | 0; 0 Long-Term Care Communities | 0; 0 Long-Term Care Communities
Period: Treatment
Arm/Group | Persons With Dementia, Experimental (LEAD IT! Programming) | Persons With Dementia, Control (Standard Care / Activity Programming)
Started | 54; 5 Long-Term Care Communities | 41; 4 Long-Term Care Communities
Completed | 51; 5 Long-Term Care Communities | 37; 4 Long-Term Care Communities
Not Completed | 3; 0 Long-Term Care Communities | 4; 0 Long-Term Care Communities
Period: Post Treatment
Arm/Group | Persons With Dementia, Experimental (LEAD IT! Programming) | Persons With Dementia, Control (Standard Care / Activity Programming)
Started | 51; 5 Long-Term Care Communities | 37; 4 Long-Term Care Communities
Completed | 47; 5 Long-Term Care Communities | 35; 4 Long-Term Care Communities
Not Completed | 4; 0 Long-Term Care Communities | 2; 0 Long-Term Care Communities

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Persons With Dementia, Experimental (LEAD IT! Programming) | Persons With Dementia, Control (Standard Care / Activity Programming) | Total
Number analyzed (Participants) | 54 | 41 | 95
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 54 | 41 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 87.13 (7.39) | 86.54 (7.06) | 86.87 (7.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 26 | 73
  Male | 7 | 15 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 54 | 41 | 95
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 1 | 8
  White | 46 | 40 | 86
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 54 | 41 | 95

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Treatment for Constructive Engagement on the Menorah Park Engagement Scale [Time Frame: Baseline (Month 1) and Treatment (Months 2, 3, and 4)
Description: Constructive Engagement on the Menorah Park Engagement Scale is defined as doing or commenting on something related to the target activity. During baseline, multiple observations of "standard" activities were observed and a single mean score was calculated for all sessions observed during that month. Then, again, during treatment, multiple treatment activity sessions were observed over the course of three months (Months 2, 3, and 4) and a single mean score was calculated. The minimum value for Constructive Engagement is zero (0) and the maximum score is two (2). Higher scores represent a better outcome.
Time Frame: Baseline (Month 1) and Treatment (Months 2, 3, and 4)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Persons With Dementia, Experimental (LEAD IT! Programming) | Persons With Dementia, Control (Standard Care / Activity Programming)
Number analyzed (Participants) | 49 | 35
score on a scale | 0.19 (0.53) | -0.24 (0.50)
Statistical Analysis 1: Comparison: Persons With Dementia, Experimental (LEAD IT! Programming) vs Persons With Dementia, Control (Standard Care / Activity Programming); Test type: Superiority; p < 0.01, ANOVA

2. Primary Outcome: Change From Baseline to Treatment for Passive Engagement on the Menorah Park Engagement Scale
Description: Passive Engagement on the Menorah Park Engagement Scale is defined as listening or watching something related to the target activity.During baseline, multiple observations of "standard" activities were observed and a single mean score was calculated for all sessions observed during that month. Then, again, during treatment, multiple treatment activity sessions were observed over the course of three months (Months 2, 3, and 4) and a single mean score was calculated. The minimum value for Passive Engagement is zero (0) and the maximum score is two (2). Higher scores represent a better outcome..
Time Frame: Baseline (Month 1) and Treatment (Months 2, 3, and 4)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Persons With Dementia, Experimental (LEAD IT! Programming) | Persons With Dementia, Control (Standard Care / Activity Programming)
Number analyzed (Participants) | 49 | 35
score on a scale | 0.69 (0.65) | -0.12 (0.55)
Statistical Analysis 1: Comparison: Persons With Dementia, Experimental (LEAD IT! Programming) vs Persons With Dementia, Control (Standard Care / Activity Programming); Test type: Superiority; p < 0.01, ANOVA

3. Primary Outcome: Change From Baseline to Treatment for Other Engagement on the Menorah Park Engagement Scale
Description: Other Engagement on the Menorah Park Engagement Scale is defined as doing, commenting, listening, or watching something NOT related to the target activity. During baseline, multiple observations of "standard" activities were observed and a single mean score was calculated for all sessions observed during that month. Then, again, during treatment, multiple treatment activity sessions were observed over the course of three months (Months 2, 3, and 4) and a single mean score was calculated. The minimum value for Other Engagement is zero (0) and the maximum score is two (2). Lower scores represent a better outcome.
Time Frame: Baseline (Month 1) and Treatment (Months 2, 3, and 4)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Persons With Dementia, Experimental (LEAD IT! Programming) | Persons With Dementia, Control (Standard Care / Activity Programming)
Number analyzed (Participants) | 49 | 35
score on a scale | -0.32 (0.48) | 0.28 (0.50)
Statistical Analysis 1: Comparison: Persons With Dementia, Experimental (LEAD IT! Programming) vs Persons With Dementia, Control (Standard Care / Activity Programming); Test type: Superiority; p < 0.01, ANOVA

4. Primary Outcome: Change From Baseline to Treatment for Non Engagement on the Menorah Park Engagement Scale
Description: Non-Engagement on the Menorah Park Engagement Scale is defined as sleeping and/or staring into space. During baseline, multiple observations of "standard" activities were observed and a single mean score was calculated for all sessions observed during that month. Then, again, during treatment, multiple treatment activity sessions were observed over the course of three months (Months 2, 3, and 4) and a single mean score was calculated. The minimum value for Non-Engagement is zero (0) and the maximum score is two (2). Lower scores represent a better outcome.
Time Frame: Baseline (Month 1) and Treatment (Months 2, 3, and 4)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Persons With Dementia, Experimental (LEAD IT! Programming) | Persons With Dementia, Control (Standard Care / Activity Programming)
Number analyzed (Participants) | 49 | 35
score on a scale | -.24 (0.35) | 0.02 (0.41)
Statistical Analysis 1: Comparison: Persons With Dementia, Experimental (LEAD IT! Programming) vs Persons With Dementia, Control (Standard Care / Activity Programming); Test type: Superiority; p < 0.01, ANOVA

5. Primary Outcome: Change From Baseline to Treatment for Pleasure on the Menorah Park Engagement Scale
Description: Pleasure on the Menorah Park Engagement Scale is defined as clearly observable laughing or smiling. During baseline, multiple observations of "standard" activities were observed and a single mean score was calculated for all sessions observed during that month. Then, again, during treatment, multiple treatment activity sessions were observed over the course of three months (Months 2, 3, and 4) and a single mean score was calculated. The minimum value for Pleasure is zero (0) and the maximum score is two (2). Lower scores represent a better outcome.
Time Frame: Baseline (Month 1) and Treatment (Months 2, 3, and 4)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Persons With Dementia, Experimental (LEAD IT! Programming) | Persons With Dementia, Control (Standard Care / Activity Programming)
Number analyzed (Participants) | 49 | 35
score on a scale | 0.32 (0.25) | -0.02 (0.27)
Statistical Analysis 1: Comparison: Persons With Dementia, Experimental (LEAD IT! Programming) vs Persons With Dementia, Control (Standard Care / Activity Programming); Test type: Superiority; p < 0.01, ANOVA

6. Secondary Outcome: Change From Baseline to Treatment on Dementia Related Quality of Life (DEMQOL)
Description: The Dementia Related Quality of Life Scale is a 28 item scale that examines quality of life in persons with dementia. The score ranges for 28 to 112. Higher scores represent a better outcome.
Time Frame: Baseline (Month 1) and Post-Treatment (Month 4)
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Persons With Dementia, Experimental (LEAD IT! Programming) | Persons With Dementia, Control (Standard Care / Activity Programming)
Number analyzed (Participants) | 47 | 34
score on scale | 1.51 (11.75) | 1.08 (15.39)
Statistical Analysis 1: Comparison: Persons With Dementia, Experimental (LEAD IT! Programming) vs Persons With Dementia, Control (Standard Care / Activity Programming); Test type: Superiority; p = 0.89, ANOVA

7. Secondary Outcome: Change From Baseline to Treatment on the Neuropsychiatric Inventory-Nursing Home (NPI-NH), Frequency x Severity Score (FxS)
Description: The NPI-NH examines 10 types of neuropsychiatric symptoms in persons with dementia, with the FxS score looking creating a composite score that takes into account frequency and severity of the symptoms. The score ranges from 0 to 120. Lower scores represent a better outcome.
Time Frame: Baseline (Month 1) and Post-Treatment (Month 4)
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Persons With Dementia, Experimental (LEAD IT! Programming) | Persons With Dementia, Control (Standard Care / Activity Programming)
Number analyzed (Participants) | 47 | 35
score on scale | -0.15 (15.32) | 3.06 (9.04)
Statistical Analysis 1: Comparison: Persons With Dementia, Experimental (LEAD IT! Programming) vs Persons With Dementia, Control (Standard Care / Activity Programming); Test type: Superiority; p = 0.27, ANOVA

8. Secondary Outcome: Change From Baseline to Treatment on the Geriatric Depression Scale-Short Form (GDS-SF)
Description: The GDS-SF consists of 15 questions requiring "yes" or "no" answers. It is specifically developed for use with older adults. For persons unable to answer the questions, a proxy can be used. The total score ranges from 0 to 15, with lower scores indicating a better outcome.
Time Frame: Baseline (Month 1) and Post-Treatment (Month 4)
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Persons With Dementia, Experimental (LEAD IT! Programming) | Persons With Dementia, Control (Standard Care / Activity Programming)
Number analyzed (Participants) | 46 | 34
score on scale | -0.71 (2.73) | 0.38 (4.58)
Statistical Analysis 1: Comparison: Persons With Dementia, Experimental (LEAD IT! Programming) vs Persons With Dementia, Control (Standard Care / Activity Programming); Test type: Superiority; p = 0.19, ANOVA

9. Secondary Outcome: Change From Baseline to Treatment on the Cohen Mansfield Agitation Inventory (CMAI)
Description: The 14-item CMAI is a caregiver rated questionnaire using a 5-point Likert scale to rate the frequency of disturbing behaviors in dementia such as verbal/physical aggression, general restlessness, strange noises, and so on. Scores range from 14 to 70, with lower scores indicating a better outcome.
Time Frame: Baseline (Month 1) and Post-Treatment (Month 4)
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Persons With Dementia, Experimental (LEAD IT! Programming) | Persons With Dementia, Control (Standard Care / Activity Programming)
Number analyzed (Participants) | 47 | 35
score on scale | -0.21 (4.53) | 2.00 (7.57)
Statistical Analysis 1: Comparison: Persons With Dementia, Experimental (LEAD IT! Programming) vs Persons With Dementia, Control (Standard Care / Activity Programming); Test type: Superiority; p = 0.10, ANOVA

ADVERSE EVENTS:
Time Frame: 5 months
Description: The communities that participated in this study were asked to report any adverse events within 48 hours of their occurrence. However, there is always a chance that they could forget to tell us about an event. So, we also do the following: once per month, a researcher contacts the key contact and asks whether any adverse events occurred in the past month. If the key contact reports an adverse event, the researcher asks for details on the event, such as date/time of occurrence, severity, etc.
Arm/Group | Persons With Dementia, Experimental (LEAD IT! Programming) | Persons With Dementia, Control (Standard Care / Activity Programming)
All-Cause Mortality (participants affected / at risk) | 2/54 | 4/41
Serious Adverse Events (participants affected / at risk) | 4/54 | 7/41
Other Adverse Events (participants affected / at risk) | 0/54 | 0/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Persons With Dementia, Experimental (LEAD IT! Programming) (N=54) | Persons With Dementia, Control (Standard Care / Activity Programming) (N=41)
Acute Illness or Injury, Sent to hospital (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Death (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-02-11): https://cdn.clinicaltrials.gov/large-docs/42/NCT05516342/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-03): https://cdn.clinicaltrials.gov/large-docs/42/NCT05516342/SAP_001.pdf